CLINICAL TRIAL: NCT02491567
Title: Study of DNA Methylation in Children and Adolescents With Autoimmune Thyroid Diseases
Brief Title: DNA Methylation and Autoimmune Thyroid Diseases
Acronym: THYRODNA
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Assimina Galli-Tsinopoulou, PROFESSOR, Aristotle University Of Thessaloniki
Other Study IDs: 62/17-2-2014
Record Dates: First submitted 2014-12-23; First posted 2015-07-08 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Hashimoto Thyroiditis; Graves Disease
MeSH Terms: conditions — Hashimoto Disease; Graves Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be collected and centrifuged and then leukocytes will be separated. DNA will then be isolated from peripheral leukocytes using the QIAamp DNA Blood Mini Kit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hashimoto Thyroiditis (HT): Children and adolescents with Hashimoto thyroiditis either hypothyroidic or euthyroidic.
- Graves Disease (GD): Children and adolescents with Graves Disease both those on remission and under antihyroid medication.
- Controls (C): Healthy individuals matched for gender and age without 1) any autoimmune disease 2) family history of autoimmune disease in the first degree relatives

SUMMARY:
Hashimoto Thyroiditis (HT) and Graves Disease (GD) are known to be caused by abnormal immune response against self cells and tissues. Epigenetics is a novel field of biology studying the mechanisms by which the environment interacts with the genotype to produce a variety of phenotypes through modifications to chromatin that do not directly alter the DNA sequence. A very limited number of epigenetic studies have been published in patients with HT and GD so far. Therefore, the purpose of this study is to analyze DNA methylation status in White Blood Cells (WBCs) within the promoter regions of genomic sites that have been previously identified as susceptibility loci or sites for autoimmune thyroid disease, such as the CD40L, FOXP3, CTLA4, PTPN22, IL2RA, FCRL3 and HLADRB1 genes.

DETAILED DESCRIPTION:
Hashimoto Thyroiditis (HT) and Graves Disease (GD) are known to be caused by abnormal immune response against self cells and tissues. HT involves a cell-mediated autoimmune destruction of the thyroid leading to hypothyroidism. GD is caused by a process in which immune cells make stimulating antibodies against the thyroid stimulating hormone (TSH) receptor on the thyroid gland, thus leading to hyperthyroidism. Although there is substantial evidence that genetic factors increase the risk for developing autoimmune diseases, monozygotic twins still remain discordant for disease (disease concordance is never 100%), thus suggesting a role for environmental factors and epigenetics.

Epigenetics is a novel field of biology studying the mechanisms by which the environment interacts with the genotype to produce a variety of phenotypes through modifications to chromatin that do not directly alter the DNA sequence. These modifications have been associated with altered gene expression and silencing of repetitive elements and can be inherited mitotically. Epigenetic mechanisms include DNA methylation, histone modifications, or miRNA post-transcriptional regulation. DNA methylation involves the covalent addition of a methyl group to the carbon-5 position in the CpG dinucleotide from the methyl donor S-adenosylmethionine and is mediated by a group of enzymes called DNA methyltransferases (DNMTs). CpG dinucleotides are typically grouped together in regions known as CGIs (islands). CGIs can be found in the promoter regions of genes, and CpG methylation of these gene promoters is associated with transcriptional silencing. In contrast, hypermethylated genes have been found to be transcriptionally active.

A very limited number of epigenetic studies have been published in patients with HT and GD so far. Therefore, the purpose of this study is to analyze DNA methylation status in White Blood Cells (WBCs) within the promoter regions of genomic sites that have been previously identified as susceptibility loci or sites for autoimmune thyroid disease, such as the CD40L, FOXP3, CTLA4, PTPN22, IL2RA, FCRL3 and HLADRB1 genes.

Initially, recruitment of patients and controls as well as blood sample collection will be done. A complete physical examination will also be performed in all participants included in the study, and a detailed personal, family, gestational and perinatal history will be obtained as well before inclusion. Blood samples by all participants will be collected and centrifuged and then White Blood Cells (WBCs), plasma and serum will be separated and stored in a deep freezer.

Laboratory analyses will follow. DNA will be isolated from peripheral leukocytes using the QIAamp DNA Blood Mini Kit, according to the manufacturer's instructions. It will then be treated with sodium bisulfite using the Zymo EZ DNA Methylation-Gold Kit, again according to the manufacturer's protocol. Therefore, unmethylated cytosines will be converted into uracyls, whereas methylated cytosines will remain unchanged. Quantification of the methylation status of DNA at the gene promoter regions under study will be made, using specific primers that detect modified DNA, by real-time PCR and analysis of the melting curves of the selected fragments of DNA. Amplicons will also be analyzed by electrophoresis and visualized by ultraviolet trans-illumination.

An electronic Data Base will be constructed and Statistical Analysis will follow. Results and Conclusions will be published in peer-review journals and presented in International Meetings.

ELIGIBILITY:
Inclusion Criteria:

For HT:

A positive titers of antithyroid peroxidase (anti-TPO) or antithyroglobulin (anti-Tg) antibodies and at least one of:

* Abnormal thyroid function that requires substitution treatment with L-thyroxine (TSH > 5 μIU/ml and decreased or normal levels of fT4 or fT3)
* Increased volume of thyroid gland (goiter)
* Morphological changes on ultrasound of the thyroid gland

For GD:

* A positive titers of thyroid stimulating antibodies (anti-TSI) and
* Decreased TSH levels and increased levels of fT4 or fT3

For Controls:

* Otherwise healthy children and adolescents, age- and gender-matched with patients
* Absence of previously known chronic disease of autoimmune aetiology or atopy (including those with a history of chronic treatment with antihistamines, anti-inflammatory, corticosteroids or anti-epileptic drugs)
* Absence of a family history of autoimmune disease in first-degree relatives

Exclusion Criteria:

* Not Caucasian origin or affinity among participants
* Age of diagnosis above 18 years
* Disease duration below 3 months

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents of Greek origin, aged 4-18 years old with a diagnosis of Hashimoto Thyroiditis and Graves Disease as well as healthy controls.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
DNA methylation status of CpGs within gene promoters | 1 month
  Percentage of DNA methylation of CpGs within the CD40L, FOXP3, CTLA4, PTPN22, IL2RA, FCRL3 and HLADRB1 promoter genes in White Blood Cells (WBCs).

SECONDARY OUTCOMES:
Age | 1 day
  Age of each participant
Age of disease onset | 1 day
  Age of disease diagnosis
Sex | 1 day
  Male or female
Body mass index | 1 day
  Weight in kg / height in m * height in m
Pubertal stage | 1 day
  Prepubertal or pubertal stage
Antibodies titre | 1 day
  Titre of antiTPO, antiTg, anti-TSI antibodies in blood
Thyroid volume | 1 day
  Volume of the thyroid gland in total (both lobes)
Treatment dose | 1 day
  Dose of Levothyroxine/thiamazole per kg of body weight /per day (if applicable)
B12 | 1 day
  Levels of B12 in blood
Folic acid | 1 day
  Levels of folic acid in blood
IgA, IgG, IgM, IgE immunoglobulins | 1 day
  Levels of IgA, IgG, IgM, IgE immunoglobulins in blood
History of infections | 1 day
  Number of previous febrile viral /bacterial infections per year
History of medications | 1 day
  Number of previous medications per year
Other autoimmune diseases | 1 day
  Diagnosis of co-existing autoimmune disease (except autoimmune thyroid disease)
Family history of autoimmune thyroid (or other) disease | 1 day
  Family history of autoimmune thyroid (or other) disease or not
Parental educational level | 1 day
  Elementary school, high school or university graduate
Type of Residence | 1 day
  Urban or rural residence
Parental smoking | 1 day
  Total number of cigarettes per day during their child's life separately for each parent (if applicable)
Previous births | 1 day
  Number of previous births
Month of birth | 1 day
  Month of birth (from January to December)
Delivery type | 1 day
  Cesarean section or vaginal delivery
Birth weight | 1 day
  Birth weight
Gestation duration | 1 day
  Duration of pregnancy
Medications during pregnancy | 1 day
  Number of medications of any type received during pregnancy (if applicable)
Maternal smoking during pregnancy | 1 day
  Total number of cigarettes per day during pregnancy (if applicable)
Maternal alcohol consumption during pregnancy | 1 day
  Total number of glasses of alcohol consumption per day during pregnancy (if applicable)
Pre-eclampsia (during pregnancy) | 1 day
  Diagnosis of pre-eclampsia (during pregnancy) or not
Gestational diabetes (during pregnancy) | 1 day
  Diagnosis of gestational diabetes (during pregnancy) or not
Vaginal bleeding (during pregnancy) | 1 day
  Presence of vaginal bleeding (during pregnancy) or not
Maternal febrile infection (during pregnancy) | 1 day
  Diagnosis of maternal febrile infection (during pregnancy) or not
Duration of breastfeeding | 1 day
  Duration of breastfeeding until discontinuance
History of phototherapy | 1 day
  History of phototherapy during neonatal period (or not)
APGAR score | 1 day
  APGAR score at 1st and 5th min of life

CONTACTS AND LOCATIONS:
Overall Officials: Assimina Galli-Tsinopoulou, Professor, Principal Investigator — Medical School, Aristotle University of Thessaloniki
Locations (1):
- Unit of Pediatric Endocrinology, Diabetes and Metabolism-4th Department of Pediatrics, Medical School of Aristotle University of Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Background] Akirav EM, Lebastchi J, Galvan EM, Henegariu O, Akirav M, Ablamunits V, Lizardi PM, Herold KC. Detection of beta cell death in diabetes using differentially methylated circulating DNA. Proc Natl Acad Sci U S A. 2011 Nov 22;108(47):19018-23. doi: 10.1073/pnas.1111008108. Epub 2011 Nov 9. PMID 22074781
- [Background] Barrett JC, Clayton DG, Concannon P, Akolkar B, Cooper JD, Erlich HA, Julier C, Morahan G, Nerup J, Nierras C, Plagnol V, Pociot F, Schuilenburg H, Smyth DJ, Stevens H, Todd JA, Walker NM, Rich SS; Type 1 Diabetes Genetics Consortium. Genome-wide association study and meta-analysis find that over 40 loci affect risk of type 1 diabetes. Nat Genet. 2009 Jun;41(6):703-7. doi: 10.1038/ng.381. Epub 2009 May 10. PMID 19430480
- [Background] Cooper JD, Simmonds MJ, Walker NM, Burren O, Brand OJ, Guo H, Wallace C, Stevens H, Coleman G; Wellcome Trust Case Control Consortium; Franklyn JA, Todd JA, Gough SC. Seven newly identified loci for autoimmune thyroid disease. Hum Mol Genet. 2012 Dec 1;21(23):5202-8. doi: 10.1093/hmg/dds357. Epub 2012 Aug 24. PMID 22922229
- [Background] Dang MN, Buzzetti R, Pozzilli P. Epigenetics in autoimmune diseases with focus on type 1 diabetes. Diabetes Metab Res Rev. 2013 Jan;29(1):8-18. doi: 10.1002/dmrr.2375. PMID 23180441
- [Background] Davies TF, Latif R, Yin X. New genetic insights from autoimmune thyroid disease. J Thyroid Res. 2012;2012:623852. doi: 10.1155/2012/623852. Epub 2012 Feb 28. PMID 22530160
- [Background] Fradin D, Le Fur S, Mille C, Naoui N, Groves C, Zelenika D, McCarthy MI, Lathrop M, Bougneres P. Association of the CpG methylation pattern of the proximal insulin gene promoter with type 1 diabetes. PLoS One. 2012;7(5):e36278. doi: 10.1371/journal.pone.0036278. Epub 2012 May 2. PMID 22567146
- [Background] Huber A, Menconi F, Corathers S, Jacobson EM, Tomer Y. Joint genetic susceptibility to type 1 diabetes and autoimmune thyroiditis: from epidemiology to mechanisms. Endocr Rev. 2008 Oct;29(6):697-725. doi: 10.1210/er.2008-0015. Epub 2008 Sep 5. PMID 18776148
- [Background] Lu Q. The critical importance of epigenetics in autoimmunity. J Autoimmun. 2013 Mar;41:1-5. doi: 10.1016/j.jaut.2013.01.010. Epub 2013 Feb 1. PMID 23375849
- [Background] MacFarlane AJ, Strom A, Scott FW. Epigenetics: deciphering how environmental factors may modify autoimmune type 1 diabetes. Mamm Genome. 2009 Sep-Oct;20(9-10):624-32. doi: 10.1007/s00335-009-9213-6. Epub 2009 Aug 22. PMID 19697079
- [Background] Quintero-Ronderos P, Montoya-Ortiz G. Epigenetics and autoimmune diseases. Autoimmune Dis. 2012;2012:593720. doi: 10.1155/2012/593720. Epub 2012 Mar 22. PMID 22536485
- [Background] Rakyan VK, Beyan H, Down TA, Hawa MI, Maslau S, Aden D, Daunay A, Busato F, Mein CA, Manfras B, Dias KR, Bell CG, Tost J, Boehm BO, Beck S, Leslie RD. Identification of type 1 diabetes-associated DNA methylation variable positions that precede disease diagnosis. PLoS Genet. 2011 Sep;7(9):e1002300. doi: 10.1371/journal.pgen.1002300. Epub 2011 Sep 29. PMID 21980303
- [Background] Weetman AP. Determinants of autoimmune thyroid disease. Nat Immunol. 2001 Sep;2(9):769-70. doi: 10.1038/ni0901-769. No abstract available. PMID 11526381
- [Background] Yin X, Latif R, Tomer Y, Davies TF. Thyroid epigenetics: X chromosome inactivation in patients with autoimmune thyroid disease. Ann N Y Acad Sci. 2007 Sep;1110:193-200. doi: 10.1196/annals.1423.021. PMID 17911434